CLINICAL TRIAL: NCT05693233
Title: Effect of Soft Robotic Exosuit Assistance in Healthy People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2022-1220
Record Dates: First submitted 2022-12-23; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Healthy Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy person (Experimental): Healthy person
  Interventions: Device: EXO On, EXO Off, EXO Removed treadmill (Uphill_incline 10°) walking and simultaneous evaluation

INTERVENTIONS:
Device: EXO On, EXO Off, EXO Removed treadmill (Uphill_incline 10°) walking and simultaneous evaluation — - After filling out the consent form for 10 subjects who meet the selection criteria, a total of three evaluations are conducted: one pre-evaluation and one post-evaluation for the knee assist robot and hip assist robot.
  Pre-evaluation: Evaluation simultaneously with walking on an inclined treadmill (Uphill_incline 10°) for 5 minutes without wearing knee and hip assist robots (speed 1.5 m/s).

SUMMARY:
This study aims to find out what effect there is on the difference in energy use efficiency and gait analysis when walking while wearing knee and hip assist robots based on flexible power structures for normal people. Energy consumption efficiency will measure the amount of energy metabolism and heart rate during walking for a set period of time, and for gait analysis, kinetic and kinematic data will be analyzed through 3D motion analysis. In addition, after completing the evaluation, we intend to help in future improvement of the product by collecting usability and satisfaction evaluation and improvements through questionnaires.

ELIGIBILITY:
Inclusion Criteria

* Healthy adults aged 19 years or older with no disabilities in walking in daily life and who have not had back or knee surgery in the past
* Those who have no problem wearing knee and hip assist robots
* A person who understands this research, has a willingness to participate voluntarily, and agrees to participate

Exclusion Criteria

- researcher judges that participation in this research is inappropriate

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
oxygen consumption measured | Simultaneous measurement of variables while walking on a treadmill_up to 24 weeks
  ① Primary evaluation variable
  - The difference between the amount of oxygen consumption measured before wearing the robot and the amount of oxygen consumption measured before and after wearing the robot [O2 rate = VO2 (ml/min) / kg of body weight, O2 cost = rate / walking speed (m/ min)].

SECONDARY OUTCOMES:
3D Motion Capture | Simultaneous measurement of variables while walking on a treadmill_up to 24 weeks
  3D Motion Capture

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol
Time Frame: Available upon request